CLINICAL TRIAL: NCT06272383
Title: Using a Single Dose of Dexamethasone at 0.6mg/kg of Body Weight Versus 0.15 mg/kg of Body Weight for the Treatment of Croup: an Internal Vanguard Randomized Controlled Non-Inferiority Trial.
Brief Title: Croup Dosing Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS26166 (B2023:092)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Results first posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Croup
Keywords: Croup, Dexamethasone, Bayesian elicitation, Dosing study, Patient engagement
MeSH Terms: conditions — Croup; Patient Participation | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is an internal double-blinded vanguard randomized controlled trial (RCT), which will be conducted at the Winnipeg Children's Hospital (WCH). Computerized randomization will be performed by a statistician at the George and Fay Yee Centre for HealthCare Innovation to generate the randomization list. Investigators will perform a computerized randomization stratified by age. Investigators will do a block randomization with random blocks of undisclosed block sizes over the seasons to ensure temporal distribution of croup cases is captured. Investigators will randomly assign patients to either the intervention or control in ratio 1:1. While croup is common between 6 months and 5 years, a typical croup affects children between 6 months and 3 years. Based on this, we will randomize such that this age category (6 months-3years) has almost similar distribution in each arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.15mg/kg dexamethasone (Experimental): Treatment with one dose of oral dexamethasone (0.15 mg/kg per dose; maximum single dose 3 mg)
  Interventions: Drug: 0.15 mg/kg dexamethasone
- Standard practice of 0.6mg/kg dexamethasone (Active Comparator): Treatment with one dose of oral dexamethasone (0.6 mg/kg per dose; maximum single dose 12 mg)
  Interventions: Drug: 0.15 mg/kg dexamethasone

INTERVENTIONS:
Drug: 0.15 mg/kg dexamethasone — 25% less than the standard practice of dexamethasone at 0.6mg/kg

SUMMARY:
Croup is a common childhood respiratory disease that often leads to frequent emergency department visits. It is a viral infection that causes cough, throat, and airway swelling, making breathing difficult. Dexamethasone is a medication that helps to reduce swelling, making breathing easier for children. A standard dose of 0.6mg/kg is used in children. However, a lower amount (due to side effects of steroids in children) has been suggested. We will examine whether 25% less than the standard dose is equally effective in treating croup. Investigators will conduct a clinical study with the support of patients with lived experience (which, in this case, are the parents of the children) to better care for children with croup. If proven, this study can improve the outcome in children with croup.

DETAILED DESCRIPTION:
Croup is a common childhood respiratory disease that leads to frequent emergency department (ED) visits. It accounts for 7% and 3% of hospitalization in under 5 and children between 6 months-3 years in North America, respectively. It is a self-limiting viral infection characterized by the sudden onset of a seal-like barking cough, often accompanied by stridor, voice hoarseness, and respiratory distress. Glucocorticoids are a class of corticosteroids with anti-inflammatory properties that help alleviate croup symptoms. While dexamethasone (a type of glucocorticoid) is commonly used to treat croup at 0.6mg/kg, a low dose of 0.15mg/kg (due to adverse events (AEs)) has been suggested to be equally effective. Investigators propose an innovative and multidisciplinary approach to investigate the noninferiority of dexamethasone at 0.15mg/kg versus 0.6mg/kg to treat croup.

ELIGIBILITY:
Inclusion Criteria:

* Children aged with clinical diagnosis of croup

Exclusion Criteria:

* Children who are unable to tolerate or ingest oral dexamethasone,
* Known hypersensitivity/allergy to dexamethasone,
* Other causes of stridor (such as acute epiglottitis, bacterial tracheitis, anaphylaxis, foreign body aspiration),
* Other underlying systemic diseases defined as chronic lung disease, chronic heart disease, chronic kidney disease, and immunodeficiency),
* Recent exposure to varicella,
* Treatment with oral or intravenous corticosteroids within the preceding 72 hours.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Aregbesola, MD, PhD, Principal Investigator — University of Manitoba; Terry Klassen, MD, MSc, Principal Investigator — University of Manitoba
Locations (1):
- Children's Hospital Winnipeg, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.15mg/kg Dexamethasone | Standard Practice of 0.6mg/kg Dexamethasone
Started | 25 | 25
Completed | 19 | 21
Not Completed | 6 | 4
Not completed — The investigational drugs were going to expire and to use the pilot data for the definitive trial | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.15mg/kg Dexamethasone | Standard Practice of 0.6mg/kg Dexamethasone | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 21 | 40
  Between 18 and 65 years | NA — Trial was conducted among children | NA — Trial was conducted among children | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Trial was conducted among children | NA — Trial was conducted among children | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 12 | 12 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight (Kg) [Mean (Full Range); unit: Kg] | 13.17 [7.50 to 18.10] | 13.69 [8.50 to 20.00] | 13.45 [7.50 to 20.00]
croup severity [Number; unit: participants] — Croup severity by Westley croup scores - mild moderate severe
  participants
    Mild croup | 16 | 16 | 32
    Moderate croup | 3 | 4 | 7
    Severe croup | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Return Visits or Readmissions to the Hospital
Description: Return visits or readmissions to the hospital within 7 days following initial presentation to the ED with croup.
Time Frame: Seven days following initial presentation to the ED with croup.
Measure: Number; unit: participants
Arm/Group | 0.15mg/kg Dexamethasone | Standard Practice of 0.6mg/kg Dexamethasone
Number analyzed (Participants) | 19 | 21
participants | 0 | 2

2. Secondary Outcome: Adverse Events
Description: Adverse events following treatment with either of the 2 doses of dexamethasone. AEs: Disseminated varicella, gastrointestinal bleeding, unspecified bleeding, pneumonia, sepsis, febrile convulsion, bacteria tracheitis, tachycardia/fast heartbeat, and restlessness.
Time Frame: within 7 and 30 days of treatment.
Measure: Number; unit: participants
Arm/Group | 0.15mg/kg Dexamethasone | Standard Practice of 0.6mg/kg Dexamethasone
Number analyzed (Participants) | 19 | 21
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: over 7 days and 30 days
Description: Patient severely ill were excluded from the study
Arm/Group | 0.15mg/kg Dexamethasone | Standard Practice of 0.6mg/kg Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT06272383/Prot_SAP_000.pdf